CLINICAL TRIAL: NCT06230029
Title: Impact of Music on Preoperative Anxiety Level Measured by Heart Rate Variability During Cataract Surgery
Brief Title: Music's Impact on Preoperative Anxiety: Heart Rate Variability Study During Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Mater Domini, Catanzaro (Other)
Responsible Party: Principal Investigator, Giuseppe Giannaccare, Professor, University of Cagliari
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Musictop2
Record Dates: First submitted 2024-01-10; First posted 2024-01-29 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Anxiety; Cataract Surgery; Heart Rate Variability
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Listening (Experimental): The presentation of the music listening session will be standardized and will be as follows: "Make yourself comfortable; we will first choose the musical style; then adjust the volume; put on the headphones; then the mask; let us know if something is wrong; we can take off the headphones or the mask at any time if you wish; we will stay by your side".
  The following data will be collected just before the headset is put on and just after its removal:
  * heart rate using a previously disinfected chest belt (PolarH10®)
  * blood pressure
  * level of anxiety (according to the validated SFQ and VAS scales)
  Music listening session will last 15 minutes, at the end of which the headphones will be removed before the patient is transferred to the operating room.
  Interventions: Other: Music listening
- No Music (No Intervention): Heart rate variability monitoring while NOT listening to music. The presentation for the patients included in the group without music will be as follows: "Make yourself comfortable; we will first put on the headphones but there will be no music; let us know if anything is wrong; we can remove the headphones or mask at any time if you wish; we will stay by your side".
  The following data will be collected just before the headset is put on and just after its removal:
  * heart rate using a previously disinfected chest belt (PolarH10®)
  * blood pressure
  * level of anxiety (according to the validated SFQ and VAS scales)
  The session will last 15 minutes, at the end of which the headphones will be removed before the patient is transferred to the operating room.

INTERVENTIONS:
Other: Music listening — Music will be played through individual headphones (BOSE AE2®). The headphones give the impression of personalized music that only the patient can hear. Patients will have a mask over their eyes to limit visual aggression. The songs will be pre-recorded on a digital tablet (Samsung Galaxy®) allowing the broadcasting of music programs. Patients will have the choice to listen to a song according to their musical preferences among 16 different musical styles. The volume will be adapted to the level that suits the patient.
  Arms: Music Listening

SUMMARY:
The goal of this Randomized Controlled Trial is to evaluate heart rate variability (HRV)before and after listening to music in patients scheduled for cataract surgery under topical anesthesia, compared to patients who do not listen to music. Our hypothesis is that the anxious population with a low HRV benefits from an anxiolytic effect of music to increase HRV levels.

ELIGIBILITY:
Inclusion Criteria:

* information and consent of the patient,
* age greater than or equal to 18 years,
* affiliation to a social security system,
* benefiting from non-emergency ambulatory cataract surgery under topical anesthesia
* not being under legal protection.

Exclusion Criteria:

* Refusal to participate,
* language barriers that are incompatible with a reliable assessment
* use of beta-blockers, including eye drops
* use of adrenergic, antiadrenergic, cholinergic and anticholinergic drugs
* use of psychotropic drugs, anxiolytics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Comparison of heart rate variability before vs after listening to music in patients scheduled for cataract surgery under topical anesthesia. | Baseline vs pre-surgery
  Use of a non-invasive sensor: recording chest belt

SECONDARY OUTCOMES:
Evaluation of the impact of music on the incidence of surgical complications | Immediately after the surgery
  Incidence of posterior capsular rupture
Measurement of subjective anxiety level | Before surgery
  Surgical Fear Questionnaire (SFQ): The questionnaire consists of 8 questions (items). The Items 1-4 refer to the subscale 'fear of short term consequences of surgery', the items 5-8 refer to the subscale 'fear of long term consequences of surgery'. All items are scored on an eleven point numeric rating scale (NRS) ranging from 0 (not at all afraid) to 10 (very afraid). This results in a total score of 0 to 80, calculated by summing item 1-8.
Measurement of subjective anxiety level | Before surgery
  Visual Analogue scale (VAS).
  In this 5-score system, we employ illustrative facial expressions to represent varying degrees of anxiety. Each segment is paired with a distinct face, visually conveying the corresponding level of anxiety:
  1. No Anxiety: The initial segment features a face showing calmness, symbolizing absence of anxiety.
  2. Mild Anxiety: The second segment depicts a face with a slightly concerned expression, indicative of mild anxiety.
  3. Moderate Anxiety: In the third segment, the face exhibits clear signs of worry, corresponding to moderate anxiety.
  4. Severe Anxiety: The fourth segment portrays a face with a deeply troubled expression, denoting severe anxiety.
  5. Extreme Anxiety: The final segment illustrates a face overwhelmed with distress, representing extreme or unbearable anxiety.
  Patients are invited to select the face that best aligns with their current perceived level of anxiety, enabling a more relatable and empathetic approach to self-assessment.

CONTACTS AND LOCATIONS:
Locations (3):
- Hôpital Cochin/Port-Royal, Paris, France
- Italy (2):
  - Eye Clinic, Department of Surgical Sciences, University of Cagliari, Cagliari
  - University of Catanzaro, Catanzaro